CLINICAL TRIAL: NCT03944018
Title: Rehabilitation Coordinators in Orthopedic Care
Acronym: REKOO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Principal Investigator, Ingrid Anderzen, associate Professor, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: REKO-O
Record Dates: First submitted 2019-05-06; First posted 2019-05-09 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2020-10

CONDITIONS: Back Problems or Pain; Foot Problems or Pain; Shoulder Problems or Pain
Keywords: Back pain
MeSH Terms: conditions — Pain; Back Pain | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention with rehabilitation coordinator (Experimental): Intervention with rehabilitation coordinator (RECO)
  Interventions: Behavioral: Intervention with rehabilitation coordinator
- Control (No Intervention): TAU

INTERVENTIONS:
Behavioral: Intervention with rehabilitation coordinator — Intervention with rehabilitation coordinator in orthopedic care
  Arms: Intervention with rehabilitation coordinator

SUMMARY:
REKO-O is a study that addressed women and men on sick leave in Uppsala County. Participants which are enrolled in orthopedic care clinic.

DETAILED DESCRIPTION:
REKO-O is a randomized controlled intervention study that addressed women and men on sick leave in Uppsala County. Participants which are enrolled in orthopedic care clinic

ELIGIBILITY:
Inclusion Criteria:

* Not recovered in accordance with care plan or cannot be operated and wants an extension of his sick leave

Exclusion Criteria:

* Obvious medical complications for surgery (wound infection, prosthetic dislocation, stopper or the like)
* Permanent disability pension

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2022-01-12 (Actual); Study Completion 2022-01-12 (Actual)

PRIMARY OUTCOMES:
RTW | 0.5 year
  Number of Participants that Return to work (RTW)

CONTACTS AND LOCATIONS:
Locations (1):
- Uppsala university, Uppsala, Sweden